CLINICAL TRIAL: NCT06061198
Title: Impact of Virtual Reality on Patient's Anxiety During Upper Limb Surgery Under Regional Anesthesia
Brief Title: Impact of Virtual Reality on Patient's Anxiety Who Underwent Surgery Uner Regional Anesthesia
Acronym: VRanxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, medical professor, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UHMahdia
Record Dates: First submitted 2023-08-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Anxiety; Satisfaction, Patient
Keywords: virtual reality; anxiety; patient satisfaction
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: 2 arms are involved in the study . first arm will receive local anesthesia with virtual reality during the surgery to reduce patient's anxiety . second arm will receive standards care under regional anesthesia
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group of patients who underwent surgery with the virtual reality experience (Active Comparator): patients underwent surgery wearing a virtual reality mask
  Interventions: Device: a virtual reality device
- patients who underwent surgery in standard conditions without the virtual reality experience (No Intervention): patients underwent surgery without a virtual reality mask

INTERVENTIONS:
Device: a virtual reality device — the patient will wear a masque tht will provide a virtual reality experience using a VR Gear connected to a mobile phone through an application installed on the mobile phone
  Arms: group of patients who underwent surgery with the virtual reality experience

SUMMARY:
this study was conducted in TAHER SFAR Hospital . it included 68 patients and it aims to evaluate the impact of virtual reality on patients undergoing upper limb surgery under regional anesthesia and evaluate the consumption of hypnotics during surgery , anxiety levels and patients satisfaction. this study contain 2 arms , each arm contain 34 patients . first arm received regional anesthesia and surgery under virtual reality using a VR gear . second arm received standard care

DETAILED DESCRIPTION:
patients who had surgery with the virtual reality experience or the VR- group ( group of patients who had surgery with standard measures without virtual reality) The patient was setup comfortably on the operating table.The echo-guided regional anesthesia appropriate to the surgical procedure is performed by an experienced anesthesiologist.In the RV+ patients, loco regional anesthesia was performed before installing the VR mask and before initiating immersing in the virtual reality space. anesthesia protocol was performed before initiating VR experience to maintain audiovisual and cognitive contact with the patient and detect possible complications For the virtual reality immersion for the VR+ group, we used an OCULUS SAMSUNG GEAR VR, a virtual reality headset connected to a SAMSUNG S7 Edge phone with headphones.The headset was worn after the loco regional anesthesia and removed at the end of the procedure.The helmet is adapted to each patient according to his head circumference measurements and the image adjustment is personalized.The VR session consists of an immersion in a natural relaxation environment produced by an application downloaded from the OCULUS STORE: VR Guided Meditation.The application offers a choice of 4 environments: Relaxing day on a tropical beach, beautiful sunset beach, mountain sunrise, or forest nap experiences . The choice of the environment is randomized according to the patient's preferences.For patients who belongs to the VR- group, the procedure was performed under standard conditions with a drape separating the patient from the operating site During surgery, the vital signs: HR, PANI, SpO2 were collected at the different peri-operative moments respectively at the entrance to the operating room (T0), 15 minutes after ALR (T1), 30 minutes after ALR (T2), 30 minutes (T3), 1 hour (T4) and 2 hours (T5) An intraoperative assessment of anxiety was performed after 15 minutes of ALR, i.e. at T1 by the LIKERT scale The anesthesist could administer anxiolytics outside of the contraindications. The molecule of choice is Midazolam and the dose taken is noted on the data collection form The administration of anxiolytics (Midazolam) is judged by clinical criteria determined in the protocol:- Anxiety during the operation judged as painful or important (higher than2 on the LIKERT scale) The session can be interrupted during the procedure for medical reasons or at the patient's request.If the local anesthesia fails and the patient is converted to general anesthesia, the protocol is cancelled and a standard induction is performed by the anesthesiologist.The events of desaturation (SpO2 < 90%), apnea, administration of anxiolytics administration of anxiolytics (to reach a minimal level of anxiety) were indicated on the data collection form.For both RV+ and RV- groups, postoperative anxiety was assessed using the scores:1- Postoperative STAI at H1 postoperative2- patient satisfaction evaluated by a LIKERT scale

ELIGIBILITY:
Inclusion Criteria:

* patient classified ASA 1 , 2 or 3
* patients undergoing an upper-limb surgery under regional anesthesia

Exclusion Criteria:

* regional anesthesia failure
* local anesthetics intoxications
* symptoms of cyber-sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
hypnovel consumption during surgery | From enrollment to the end of treatment at 10 weeks
  the required dose of Midazolam for a LIKERT intraoperative anxiety score goal < 2

SECONDARY OUTCOMES:
satisfaction level during surgery | at the end of the procedure
  satisfaction levels measured with a LIKERT scale : 1 : not satisfied , 2: low satisfaction , 3:satisfied , 4: great satisfaction
pre-operative patients's anxiety level by LIKERT score | From enrollment to the end of treatment at 10 weeks
  pre operative anxiety measured with a LIKERT scale : 1= no anxiety , 2: tolerable anxiety , 3= anxious ; 4= hard experience
per-operative patients's anxiety level by LIKERT score | From enrollment to the end of treatment at 10 weeks
  per operative anxiety measured with a LIKERT scale : 1= no anxiety , 2: tolerable anxiety , 3= anxious ; 4= hard experience
post-operative patients's anxiety level by LIKERT score | From enrollment to the end of treatment at 10 weeks
  post operative anxiety measured with a LIKERT scale: 1= no anxiety , 2: tolerable anxiety , 3= anxious ; 4= hard experience
vitals : systolic pressure | From enrollment to the end of treatment at 10 weeks
  vitals were monitored all long the procedure
vitals : heart rate | From enrollment to the end of treatment at 10 weeks
  vitals were monitored all long the procedure
vitals : oxygen saturation | From enrollment to the end of treatment at 10 weeks
  vitals were monitored all long the procedure
pre-operative patients's anxiety level by STAI-6 score | From enrollment to the end of treatment at 10 weeks
  pre operative anxiety measured with a STAI-6 modified scale : a total score superior to 65 : high anxiety , score between 56-65 : too high anxiety , score between : 36 - 45 : low anxiety , score inferior to 35 no anxiety
post-operative patients's anxiety level by STAI-6 score | From enrollment to the end of treatment at 10 weeks
  post operative anxiety measured with a STAI-6 modified scale : a total score superior to 65 : high anxiety , score between 56-65 : too high anxiety , score between : 36 - 45 : low anxiety , score inferior to 35 no anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Majdoub Ali MD, professor, Principal Investigator — University Hospital, Mahdia
Locations (1):
- Taher Sfar University Hospital, Mahdia, Tunisia

IPD SHARING:
Plan to Share IPD: No